CLINICAL TRIAL: NCT03532620
Title: A Multi-center, Open-label, Randomized, 12-month, Parallel-group, Non-inferiority Study to Compare the Hemoglobin A1C Metabolism of Pitavastatin Therapy Versus Atorvastatin in Chinese Patients With Prediabetes and Hypertension
Brief Title: China Protection Trial of Glucose Metabolism by Pitavastatin in Patients With Prediabetes and Hypertension
Acronym: CAMPUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun Tao (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Jun Tao, Director, Head of the Department of Hypertension and Cardiovascular Disease, Principal Investigator, Clinical Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BZ-1702
Record Dates: First submitted 2018-04-27; First posted 2018-05-22 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Prediabetic State; Hypertension; Dyslipidemias
Keywords: Pitavastatin; Prediabetic State; Hypertension; Dyslipidemias; Cardiovascular Disease
MeSH Terms: conditions — Prediabetic State; Hypertension; Dyslipidemias; Cardiovascular Diseases | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- pitavastatin (Experimental): Pitavastatin Calcium + lifestyle modification
  Interventions: Drug: Pitavastatin Calcium
- atorvastatin (Active Comparator): Atorvastatin Calcium + lifestyle modification
  Interventions: Drug: Atorvastatin Calcium

INTERVENTIONS:
Drug: Pitavastatin Calcium — In Pitavastatin treatment group, Pitavastatin calcium tablet 2mg/day was given for 12 months in combination with lifestyle modification. But month 3 is the "check point". If LDL-C target was achieved at Month 3, doses remained the same. If LDL-C target was not achieved at Month 3, doses were doubled.
  Arms: pitavastatin
Drug: Atorvastatin Calcium — In Atorvastatin treatment group, Atorvastatin calcium tablet 20mg/day was given for 12 months in combination with lifestyle modification. But month 3 is the "check point". If LDL-C target was achieved at Month 3, doses remained the same. If LDL-C target was not achieved at Month 3, doses were doubled.
  Other Names: Lipitor®
  Arms: atorvastatin

SUMMARY:
The primary purpose of this trial is to test the hypothesis that Pitavastatin treatment compared to Atorvastatin, in patients with dyslipidemia, prediabetes and hypertension, will have less adverse effect on Hemoglobin A1C (HbA1C), which represents long-term glucose metabolism.

DETAILED DESCRIPTION:
Within the 12 months of the study procedure, the 3rd month is what we called the "check point". At this point, participants' plasma LDL-C will be measured whether it reached individual standard or not. If the results didn't meet the particular LDL-C standard, the participants would be adjusted the drug dosage (pitavastatin 4mg/day, atorvastatin 40mg/day).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. IFG: 5.6mmol/L (100mg/dl)≤FPG<7.0mmol/L (126mg/dl), or IGT: 7.8mmol/L (140mg/dl)≤OGTT 2-h PG<11.1mmol/L (200mg/dl), or HbA1C 5.7-6.4% (39-47mmol/mol);
3. 2.6mmol/L (100mg/dl)≤LDL-C≤5.2mmol/L (200mg/dl), and TG<5.7mmol/L (500mg/dl);
4. 130mmHg≤SBP<180mmHg, or 80mmHg≤DBP<110mmHg or ongoing anti-hypertensive therapy;
5. Patients volunteered for the study and signed informed consent.

Exclusion Criteria:

1. Past history of hypersensitivity to the study drug;
2. Diagnosed diabetes;
3. Severe liver disease (including ALT or AST≥2.5-fold the normal upper limit), biliary obstruction;
4. Ongoing treatment with cyclosporine within 2 weeks;
5. Renal dysfunction, including endogenous creatinine clearance male<120ml/min, female<105ml/min, serum creatinine≥2mg/dl (186umol/L), Renal function progressive decline, GFR<30ml•min-1•1.73m-2;
6. Diagnosed or past history of ASCVD (including ACS, SCAD, revascularization, ICM, ischemic stroke, TIA, PASD, etc.
7. SBP≥180mmHg, or DBP≥110mmHg;
8. Ongoing treatment with Beta blockers, Diuretic;
9. Secondary hypertension, including SAS, PA, RAS, pheochromocytoma, Cushing's syndrome, aorta diseases, drug induced hypertension;
10. Ongoing treatment with statins, fibrates, and/or cation exchange resins within 2 weeks;
11. Pancreatic disease;
12. History of gastrectomy, short bowel syndrome;
13. Ongoing hormone replacement therapy;
14. Diagnosed or suspected malignant tumor;
15. Familial hypercholesterolemia;
16. Any diseases may limit the efficacy or safety of the study;
17. Pregnant or possibly pregnant woman, or breastfeeding woman, or woman who wishes to become pregnant during study participation;
18. Patient who was not judged as eligible by the investigator/coinvestigator.

    * IFG impaired fast glucose, FPG fasting plasma glucose, IGT impaired glucose tolerance, OGTT oral glucose tolerance test, PG plasma glucose, HbA1C hemoglobin A1C, LDL-C low-density lipoprotein cholesterol, TG triglycerides, SBP systolic blood pressure, DBP diastolic blood pressure, ALT alanine aminotransferase, AST aspartate aminotransferase, GFR glomerular filtration rate, ASCVD arteriosclerotic cardiovascular disease, ACS acute coronary syndrome, SCAD stable coronary artery disease, ICM ischemic cardiomyopathy, TIA transient ischemic attack, PASD peripheral atherosclerotic disease, SAS sleep apnea syndrome, PA primary aldosteronism, RAS renal arterial stenosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin A1c levels | Month 12
  Change of HbA1C values at study initiation and study completion

SECONDARY OUTCOMES:
Changes from baseline in FPG levels | Month 12
  Change of fasting plasma glucose (FPG) values at study initiation and study completion
Changes from baseline in OGTT-2h PG levels | Month 12
  Change of oral glucose tolerance test (OGTT)-2h plasma glucose (PG) values at study initiation and study completion
Proportion of subjects in LDL-C normalization state | Month 3 and 12
  Proportion of subjects in each group who achieved low-density lipoprotein cholesterol (LDL-C) target
Changes from baseline in high-density lipoprotein cholesterol (HDL-C) levels | Month 12
  Change of HDL-C values at study initiation and study completion
Changes from baseline in total cholesterol (TC) levels | Month 12
  Change of TC values at study initiation and study completion
Changes from baseline in triglycerides (TG) levels | Month 12
  Change of TG values at study initiation and study completion
Changes from baseline in inflammatory parameters | Month 12
  Change of C-reactive protein (CRP) values at study initiation and study completion
Incidence of cardiovascular disease (CVD) events | Month 12
  Incidence of cardiovascular disease (CVD) events, including acute coronary syndrome, stable coronary artery disease, ischemic cardiomyopathy etc.
Change from baseline in blood pressure levels | Month 12
  Change from baseline in systolic and diastolic blood pressure levels
Changes from baseline in vascular endothelial function | Month 12
  Change of brachial-ankle pulse wave velocity (baPWV) values at study initiation and study completion
Changes from baseline in left ventricular mass index | Month 12
  Change of left ventricular mass index (LVMI) values at study initiation and study completion
Changes from baseline in carotid intima-media thickness | Month 12
  Change of carotid intima-media thickness (CIMT) values at study initiation and study completion

OTHER OUTCOMES:
Incidence of adverse events (AEs) | Month 12
  Incidence of adverse events (AEs) after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Jun Tao, MD,PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (13):
- China (13):
  - Fourth People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - People's Hospital of Zhongshan City, Zhongshan, Guangdong
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, He'nan
  - Yichang Central Hospital, Yichang, Hubei
  - Taizhou Hospital of TCM, Taizhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - Lanzhou University Second Hospital, Lanzhou, Qinghai
  - Yantaishan Hospital, Yantai, Yantai, Shandong

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, Statistical Analysis Plan, Clinical Study Report are planned to be available to other researchers. The information will be published on scientific journal and is anticipated to be available in public no more than a year after the study completion.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Study protocol will be published on scientific journal and is anticipated to be available online by the end of 2018. Statistical Analysis Plan will be finished before the trial ends. Clinical Study Report will be published in public no more than a year after the study completion.
Access Criteria: All researchers will be available to get the individual participant data (IPD) as long as the information is published.

REFERENCES:
- [Background] Maki KC, Ridker PM, Brown WV, Grundy SM, Sattar N, The Diabetes Subpanel of the National Lipid Association Expert Panel. An assessment by the Statin Diabetes Safety Task Force: 2014 update. J Clin Lipidol. 2014 May-Jun;8(3 Suppl):S17-29. doi: 10.1016/j.jacl.2014.02.012. PMID 24793439
- [Background] Yusuf S, Lonn E, Pais P, Bosch J, Lopez-Jaramillo P, Zhu J, Xavier D, Avezum A, Leiter LA, Piegas LS, Parkhomenko A, Keltai M, Keltai K, Sliwa K, Chazova I, Peters RJ, Held C, Yusoff K, Lewis BS, Jansky P, Khunti K, Toff WD, Reid CM, Varigos J, Accini JL, McKelvie R, Pogue J, Jung H, Liu L, Diaz R, Dans A, Dagenais G; HOPE-3 Investigators. Blood-Pressure and Cholesterol Lowering in Persons without Cardiovascular Disease. N Engl J Med. 2016 May 26;374(21):2032-43. doi: 10.1056/NEJMoa1600177. Epub 2016 Apr 2. PMID 27039945
- [Background] Baudrand R, Pojoga LH, Vaidya A, Garza AE, Vohringer PA, Jeunemaitre X, Hopkins PN, Yao TM, Williams J, Adler GK, Williams GH. Statin Use and Adrenal Aldosterone Production in Hypertensive and Diabetic Subjects. Circulation. 2015 Nov 10;132(19):1825-33. doi: 10.1161/CIRCULATIONAHA.115.016759. Epub 2015 Oct 2. PMID 26432671
- [Background] Warita S, Kawasaki M, Tanaka R, Ono K, Kojima T, Hirose T, Iwama M, Watanabe T, Nishigaki K, Takemura G, Noda T, Watanabe S, Minatoguchi S. Effects of pitavastatin on cardiac structure and function and on prevention of atrial fibrillation in elderly hypertensive patients: a prospective study of 2-years' follow-up. Circ J. 2012;76(12):2755-62. doi: 10.1253/circj.cj-12-0722. Epub 2012 Aug 8. PMID 22878405
- [Background] Yoshika M, Komiyama Y, Masuda M, Yokoi T, Masaki H, Ohkura H, Takahashi H. Pitavastatin further decreases serum high-sensitive C-reactive protein levels in hypertensive patients with hypercholesterolemia treated with angiotensin II, type-1 receptor antagonists. Clin Exp Hypertens. 2010;32(6):341-6. doi: 10.3109/10641961003628460. PMID 21028996
- [Background] Pearson TA, Mensah GA, Alexander RW, Anderson JL, Cannon RO 3rd, Criqui M, Fadl YY, Fortmann SP, Hong Y, Myers GL, Rifai N, Smith SC Jr, Taubert K, Tracy RP, Vinicor F; Centers for Disease Control and Prevention; American Heart Association. Markers of inflammation and cardiovascular disease: application to clinical and public health practice: A statement for healthcare professionals from the Centers for Disease Control and Prevention and the American Heart Association. Circulation. 2003 Jan 28;107(3):499-511. doi: 10.1161/01.cir.0000052939.59093.45. No abstract available. PMID 12551878
- [Background] Kushiro T, Mizuno K, Nakaya N, Ohashi Y, Tajima N, Teramoto T, Uchiyama S, Nakamura H; Management of Elevated Cholesterol in the Primary Prevention Group of Adult Japanese Study Group. Pravastatin for cardiovascular event primary prevention in patients with mild-to-moderate hypertension in the Management of Elevated Cholesterol in the Primary Prevention Group of Adult Japanese (MEGA) Study. Hypertension. 2009 Feb;53(2):135-41. doi: 10.1161/HYPERTENSIONAHA.108.120584. Epub 2008 Dec 22. PMID 19104004
- [Background] Ridker PM, Danielson E, Fonseca FA, Genest J, Gotto AM Jr, Kastelein JJ, Koenig W, Libby P, Lorenzatti AJ, MacFadyen JG, Nordestgaard BG, Shepherd J, Willerson JT, Glynn RJ; JUPITER Study Group. Rosuvastatin to prevent vascular events in men and women with elevated C-reactive protein. N Engl J Med. 2008 Nov 20;359(21):2195-207. doi: 10.1056/NEJMoa0807646. Epub 2008 Nov 9. PMID 18997196
- [Background] Ridker PM, Macfadyen JG, Nordestgaard BG, Koenig W, Kastelein JJ, Genest J, Glynn RJ. Rosuvastatin for primary prevention among individuals with elevated high-sensitivity c-reactive protein and 5% to 10% and 10% to 20% 10-year risk. Implications of the Justification for Use of Statins in Prevention: an Intervention Trial Evaluating Rosuvastatin (JUPITER) trial for "intermediate risk". Circ Cardiovasc Qual Outcomes. 2010 Sep;3(5):447-52. doi: 10.1161/CIRCOUTCOMES.110.938118. Epub 2010 Aug 24. PMID 20736443
- [Derived] Zhang J, Shao Y, Liu Y, Tao J. A Multi-Center, Open-Label, Two-Arm Parallel Group Non-inferiority Randomized Controlled Trial Evaluating the Effect of Pitavastatin, Compared to Atorvastatin, on Glucose Metabolism in Prediabetics with Hypertension and Dyslipidemia: Rationale and Design for the China Hemoglobin A1c Metabolism Protection Union Study (CAMPUS). Cardiovasc Drugs Ther. 2018 Dec;32(6):581-589. doi: 10.1007/s10557-018-6826-6. PMID 30187345